CLINICAL TRIAL: NCT00069641
Title: A Phase II/III, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety and Efficacy of Weekly and Every Other Week Dosing Regimens of Iduronate-2-Sulfatase Enzyme Replacement Therapy in Patients With MPS II
Brief Title: Iduronate-2-sulfatase Enzyme Replacement Therapy in Mucopolysaccharidosis II (MPS II)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TKT024
Record Dates: First submitted 2003-09-29; First posted 2003-10-01 (Estimated); Results first posted 2015-05-13 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Mucopolysaccharidosis II
Keywords: Mucopolysaccharidosis II; MPS II; Hunter Syndrome; iduronate-2-sulfatase; I2S; Iduronate-2-sulfatase deficiency
MeSH Terms: conditions — Mucopolysaccharidosis II; Sudden Infant Death | interventions — idursulfase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Idursulfase weekly (0.5 mg/kg) (Experimental)
  Interventions: Biological: Iduronate-2-sulfatase enzyme replacement therapy
- Idursulfase every other week (0.5 mg/kg) (Experimental)
  Interventions: Biological: iduronate-2-sulfatase enzyme replacement therapy
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Iduronate-2-sulfatase enzyme replacement therapy — Patients will receive weekly infusions of idursulfase at a dose of 0.5 mg/kg.
  Other Names: Elaprase
  Arms: Idursulfase weekly (0.5 mg/kg)
Biological: iduronate-2-sulfatase enzyme replacement therapy — Patients will receive every other week infusions of idursulfase at a dose of 0.5 mg/kg.
  Other Names: Elaprase
  Arms: Idursulfase every other week (0.5 mg/kg)
Biological: Placebo — Patients will receive weekly infusions of placebo.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether the administration of iduronate-2-sulfatase enzyme in a weekly or every other week therapy frequency is safe and efficacious in patients with MPS II.

DETAILED DESCRIPTION:
MPS II is a rare, X-linked, lysosomal storage disorder caused by a deficiency in the enzyme iduronate-2-sulfatase. Because of this deficiency, glycosaminoglycans (GAG) accumulate in multiple tissues and organs, resulting in progressive cellular and organ system dysfunction. The purpose of this study is to determine if one year of therapy with iduronate-2-sulfatase enzyme replacement therapy, at a dose of 0.5mg/kg, weekly or every other week, is safe, and results in clinically meaningful improvement in multiple organ function, compared with a placebo group. Upon completion of the study, patients will be eligible to enroll in an open-label maintenance study.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, patients must meet the following inclusion criteria prior to enrollment:

1. The diagnosis of MPS II will be determined by the investigator based upon both clinical and biochemical criteria.
2. All patients must have at least one of the following Clinical Criteria considered by the investigator to be MPS II-related:

   * Hepatosplenomegaly
   * Radiographic evidence of dysostosis multiplex
   * Valvular heart disease
   * Evidence of obstructive pulmonary disease
3. In addition, patients must have the following Biochemical Criteria:

   * Documented deficiency in iduronate-2-sulfastase enzyme activity of less than or equal to 10% of the lower limit of the normal range as measured in plasma, fibroblasts, or leukocytes (based on normal range of measuring laboratory).
   * A normal enzyme activity level of one other sulfatase as measured in plasma, fibroblasts, or leukocytes (based on normal range of measuring laboratory).
4. Must be male, 5 to 25 years of age.
5. Forced vital capacity of <80% of predicted obtained at the baseline evaluation of this study.
6. Must be able to adequately perform the testing required in this study, including reproducible pulmonary function testing by spirometry, as judged by the investigator.
7. Patient, patient's parent(s), or legally authorized guardian must have voluntarily signed an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved informed consent form after all relevant aspects of the study have been explained and discussed with the patient.

Exclusion Criteria:

Patients meeting any of the following criteria are not eligible for participation in this study:

1. Patient has received treatment with another investigational therapy within the past 60 days.
2. Patient, patient's parent(s), or patient's legal guardian is unable to understand the nature, scope, and possible consequences of the study.
3. Patient is unable to comply with the protocol (e.g., due to a medical condition such as cervical cord compression or uncooperative attitude) or is unlikely to complete the study, as determined by the investigator.
4. Patient has a tracheostomy.
5. Patient has received a bone marrow or cord blood transplant.
6. Patient with known hypersensitivity to any of the components of iduronate-2-sulfatase.

Ages: 5 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 96 (Actual)
Dates: Start 2003-09-18 (Actual); Primary Completion 2005-03-16 (Actual); Study Completion 2005-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (9):
- United States (4):
  - Children's Hospital Oakland, Oakland, California
  - St. Louis Children's Hospital, Washington University, St Louis, Missouri
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Texas Children's Hospital, Baylor College of Medicine, Houston, Texas
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Brazil
- Children's Hospital, Johannes-Gutenburg Universitaet Mainz, Mainz, Germany
- United Kingdom (3):
  - Addenbrooke's Hospital, Cambridge, England
  - Great Ormond Street Hospital for Sick Children, London, England
  - Royal Manchester Children's Hospital, Manchester, England

REFERENCES:
- [Derived] Tandon PK, Kakkis ED. The multi-domain responder index: a novel analysis tool to capture a broader assessment of clinical benefit in heterogeneous complex rare diseases. Orphanet J Rare Dis. 2021 Apr 19;16(1):183. doi: 10.1186/s13023-021-01805-5. PMID 33874971
- [Derived] Raluy-Callado M, Chen WH, Whiteman DA, Fang J, Wiklund I. The impact of Hunter syndrome (mucopolysaccharidosis type II) on health-related quality of life. Orphanet J Rare Dis. 2013 Jul 10;8:101. doi: 10.1186/1750-1172-8-101. PMID 23837440

RESULTS

PARTICIPANT FLOW:
Groups:
- Idursulfase Weekly (0.5 mg/kg): Idursulfase 0.5 milligram per kilogram (mg/kg) administered once-weekly by intravenous infusion for one year (52 infusions).
- Idursulfase Every Other Week (EOW) (0.5 mg/kg): Idursulfase 0.5 mg/kg administered every other week by intravenous infusion for one year (26 infusions) along with placebo matching to idursulfase every other week (alternating with idursulfase) by intravenous infusion for one year (26 infusions).
- Placebo: Placebo matching to idursulfase administered once-weekly by intravenous infusion for one year (52 infusions).
Period: Overall Study
Arm/Group | Idursulfase Weekly (0.5 mg/kg) | Idursulfase Every Other Week (EOW) (0.5 mg/kg) | Placebo
Started | 32 | 32 | 32
Completed | 31 | 32 | 31
Not Completed | 1 | 0 | 1
Not completed — Death | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Idursulfase Weekly (0.5 mg/kg): Idursulfase 0.5 mg/kg administered once-weekly by intravenous infusion for one year (52 infusions).
- Idursulfase EOW (0.5 mg/kg): Idursulfase 0.5 mg/kg administered every other week by intravenous infusion for one year (26 infusions) along with placebo matching to idursulfase every other week (alternating with idursulfase) by intravenous infusion for one year (26 infusions).
- Total: Total of all reporting groups
Arm/Group | Idursulfase Weekly (0.5 mg/kg) | Idursulfase EOW (0.5 mg/kg) | Placebo | Total
Number analyzed (Participants) | 32 | 32 | 32 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at randomization.
  years | 15.14 (6.293) | 14.40 (7.019) | 13.12 (6.908) | 14.22 (6.729)
Age, Customized [Count of Participants; unit: Participants] — Age at randomization. The participant who was less than (<) 5 years old was considered for randomization to be in 5 to 11 years category. Participants who were greater than (>) 25 years old were considered for randomization to be in 19 to 25 years category.
  Participants
    5 to 11 years | 14 | 14 | 15 | 43
    12 to 18 years | 10 | 9 | 10 | 29
    19 to 25 years | 7 | 7 | 5 | 19
    greater than equal to (>=) 26 years | 1 | 2 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 32 | 32 | 32 | 96
Region of Enrollment [Count of Participants; unit: Participants]
  North America | 11 | 11 | 12 | 34
  South America | 7 | 7 | 7 | 21
  Europe | 14 | 14 | 13 | 41

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in Mean Global Joint Range of Motion (JROM) Score at Week 53
Description: Change was calculated at Week 53 from baseline. Global JROM (% of normal range of motion) is the average of 11 ratios multiplied by 100. Ratios are Left/Right means of passive range of motion in Shoulder (Flexion/Extension, Abduction, Internal/External Rotation), Elbow (Flexion/Extension), Wrist (Flexion/Extension), Index Finger (Flexion/Extension [Combined Metacarpophalangeal joint (MCP), Proximal interphalangeal joint (PIP), Distal interphalangeal joint (DIP) motion]), Hip (Flexion/Extension, Abduction, Internal/External Rotation), Knee (Flexion/Extension), and Ankle (Dorsiflexion) divided by the normal range (American Academy of Orthopedic Surgeons and American Medical Association).
Time Frame: Baseline, Week 53
Population: ITT population. Here, number of participants analyzed = participants who were evaluable for this measure.
Measure: Mean (Standard Error); unit: percentage of normal range of motion
Arm/Group | Idursulfase Weekly (0.5 mg/kg) | Idursulfase EOW (0.5 mg/kg) | Placebo
Number analyzed (Participants) | 31 | 32 | 31
percentage of normal range of motion
  Baseline | 66.86 (1.85) | 67.36 (1.43) | 67.70 (1.59)
  Change at Week 53 | 0.89 (0.87) | -0.61 (0.94) | 0.70 (1.10)

2. Secondary Outcome: Mean Combined Liver and Spleen Volume at Baseline
Description: Liver and Spleen volume was determined by Magnetic Resonance Imaging (MRI).
Time Frame: Baseline
Population: ITT population. Here, number of participants analyzed = participants who were evaluable for this measure.
Measure: Mean (Standard Error); unit: milliliter (mL)
Arm/Group | Idursulfase Weekly (0.5 mg/kg) | Idursulfase EOW (0.5 mg/kg) | Placebo
Number analyzed (Participants) | 31 | 29 | 30
milliliter (mL) | 1578.48 (80.75) | 1442.2 (63.54) | 1485.28 (70.19)

3. Secondary Outcome: Percent Change From Baseline in Mean Combined Liver and Spleen Volume at Week 53
Description: Liver and Spleen volume was determined by Magnetic Resonance Imaging (MRI). Change was calculated at Week 53 from baseline.
Time Frame: Baseline, Week 53
Population: ITT population. Here, number of participants analyzed = participants who were evaluable for this measure.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Idursulfase Weekly (0.5 mg/kg) | Idursulfase EOW (0.5 mg/kg) | Placebo
Number analyzed (Participants) | 31 | 29 | 30
percent change | -25.81 (1.44) | -23.73 (1.49) | 0.27 (1.66)

4. Secondary Outcome: Change From Baseline in Mean Normalized Urine Glycosaminoglycan (GAG) Levels at Week 53
Description: Mean normalized urine GAG was analyzed using urine testing. Change was calculated at Week 53 from baseline. The urine GAG levels were normalized to urine creatinine and were reported as microgram GAG per milligram creatinine (mcg GAG/mg creatinine).
Time Frame: Baseline, Week 53
Population: ITT population.
Measure: Mean (Standard Error); unit: mcg GAG/mg creatinine
Arm/Group | Idursulfase Weekly (0.5 mg/kg) | Idursulfase EOW (0.5 mg/kg) | Placebo
Number analyzed (Participants) | 32 | 32 | 32
mcg GAG/mg creatinine
  Baseline | 325.59 (25.79) | 338.08 (21.03) | 419.40 (34.37)
  Change at Week 53 | -189.23 (25.76) | -154.98 (17.18) | 18.16 (29.94)

5. Primary Outcome: Ranked Adjusted 2-Component Composite Variable Score Based on Change From Baseline to Week 53
Description: The 2-component composite variable consists of the sum of the ranked changes from baseline to Week 53 for percent predicted Forced Vital Capacity (FVC) and 6-Minute Walking Test (6MWT) total distance walked. For the 2 treatment groups being compared, ranking occurred within the comparison treatment groups combined (idursulfase weekly and placebo treatment groups). These comparison groups were pooled and ranked for each component separately. Within each component (% predicted FVC, 6MWT), the change from baseline was then ranked. The lowest change value was assigned a rank of 1, the next lowest a rank of 2, etc. The composite score for each participant was the sum of the 2 ranked scores corresponding to the 2 individual components (% predicted FVC and 6MWT) for each participant. Thus, the greater the composite score (greater the sum of the ranks of the changes from baseline, where the lowest change was ranked as 1), the greater the improvement.
Time Frame: Baseline, Week 53
Population: Intent-to-treat (ITT) population, Only participants receiving "Idursulfase Weekly" or "Placebo" were to be analyzed for this outcome.
Measure: Mean (Standard Error); unit: sum of the ranked scores
Arm/Group | Idursulfase Weekly (0.5 mg/kg) | Placebo
Number analyzed (Participants) | 32 | 32
sum of the ranked scores | 69.81 (7.03) | 50.86 (8.07)
Statistical Analysis 1: Comparison: Idursulfase Weekly (0.5 mg/kg) vs Placebo; p-value for treatment difference based on Analysis of covariance (ANCOVA) model containing treatment, region, baseline participant age, and baseline disease score; Test type: Superiority or Other; p = 0.0049, ANCOVA; Mean Difference (Net) = 18.96, 95% CI 2-sided [5.99 to 31.93], Standard Error of Mean 6.47

6. Secondary Outcome: Mean Cardiac Left Ventricular Mass Index (LVMI) at Baseline
Description: Cardiac LVMI was determined by echocardiography. LVMI is the left ventricular mass (LVM, in grams [g]) indexed to body surface area (BSA), in square meter [m^2]. LVMI (in gram per square meter [g/m^2]) = LVM divided by BSA.
Time Frame: Baseline
Population: ITT population. Here, number of participants analyzed = participants who were evaluable for this measure.
Measure: Mean (Standard Error); unit: gram per square meter (g/m^2)
Arm/Group | Idursulfase Weekly (0.5 mg/kg) | Idursulfase EOW (0.5 mg/kg) | Placebo
Number analyzed (Participants) | 31 | 31 | 31
gram per square meter (g/m^2) | 105.18 (6.86) | 89.42 (4.38) | 95.55 (5.96)

7. Secondary Outcome: Percent Change From Baseline in Mean Cardiac Left Ventricular Mass Index (LVMI) at Week 53
Description: Cardiac LVMI was determined by echocardiography. Change was calculated at Week 53 from baseline. LVMI is the LVM, in grams indexed to BSA, in square meter [m^2]. LVMI in g/m^2 = LVM divided by BSA.
Time Frame: Baseline, Week 53
Population: ITT population. Here, number of participants analyzed = participants who were evaluable for this measure.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Idursulfase Weekly (0.5 mg/kg) | Idursulfase EOW (0.5 mg/kg) | Placebo
Number analyzed (Participants) | 31 | 31 | 31
percent change | -1.34 (5.05) | 6.71 (4.03) | 3.56 (4.12)

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Idursulfase Weekly (0.5 mg/kg) | Idursulfase EOW (0.5 mg/kg) | Placebo
Serious Adverse Events (participants affected / at risk) | 9/32 | 8/32 | 9/32
Other Adverse Events (participants affected / at risk) | 32/32 | 32/32 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Idursulfase Weekly (0.5 mg/kg) (N=32) | Idursulfase EOW (0.5 mg/kg) (N=32) | Placebo (N=32)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Arrhythmia not otherwise specified (nos) (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cyanosis nos (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Heart valve insufficiency (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ear disorder nos (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Otorrhoea (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia nos (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hernia nos (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchopneumonia nos (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis media chronic nos (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Otitis media serous nos (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pilonidal sinus infected (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth caries nos (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound infection due to staphylococcus aureus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Anaesthesia intubation complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Medical device complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood carbon dioxide increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Phobia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm nos (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rash nos (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Poor venous access (Vascular disorders) | 2 (2) | 3 (4) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Idursulfase Weekly (0.5 mg/kg) (N=32) | Idursulfase EOW (0.5 mg/kg) (N=32) | Placebo (N=32)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Atrial hypertrophy (Cardiac disorders) | 2 (2) | 0 (0) | 3 (3)
Tachycardia nos (Cardiac disorders) | 1 (1) | 3 (5) | 2 (10)
Ventricular hypertrophy (Cardiac disorders) | 2 (2) | 2 (2) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 2 (2)
Deafness nos (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 2 (2)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
Ear disorder nos (Ear and labyrinth disorders) | 2 (3) | 1 (1) | 0 (0)
Ear haemorrhage (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (3)
Ear pain (Ear and labyrinth disorders) | 7 (7) | 5 (9) | 6 (13)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 (1) | 2 (5) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 5 (5) | 4 (5)
Otorrhoea (Ear and labyrinth disorders) | 7 (20) | 7 (17) | 9 (21)
Sensation of block in ear (Ear and labyrinth disorders) | 0 (0) | 3 (3) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 3 (3)
Conjunctivitis allergic (Eye disorders) | 2 (2) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 3 (3) | 1 (1) | 1 (1)
Hypermetropia (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 3 (6) | 0 (0) | 1 (2)
Myopia (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Vision blurred (Eye disorders) | 3 (5) | 0 (0) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Abdominal pain nos (Gastrointestinal disorders) | 11 (24) | 17 (36) | 11 (20)
Abdominal pain upper (Gastrointestinal disorders) | 5 (14) | 2 (2) | 2 (3)
Constipation (Gastrointestinal disorders) | 2 (4) | 1 (1) | 1 (2)
Diarrhoea nos (Gastrointestinal disorders) | 11 (22) | 12 (24) | 15 (29)
Dyspepsia (Gastrointestinal disorders) | 4 (5) | 4 (18) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (13) | 1 (1)
Gastroenteritis nos (Gastrointestinal disorders) | 1 (1) | 3 (4) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Inguinal hernia nos (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Loose stools (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (4)
Nausea (Gastrointestinal disorders) | 7 (18) | 9 (16) | 9 (17)
Swollen tongue (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Umbilical hernia nos (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Vomiting nos (Gastrointestinal disorders) | 8 (22) | 18 (37) | 16 (43)
Asthenia (General disorders) | 3 (3) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 2 (3) | 3 (3)
Chest pain (General disorders) | 3 (7) | 2 (2) | 0 (0)
Fall (General disorders) | 0 (0) | 4 (7) | 4 (10)
Fatigue (General disorders) | 2 (2) | 4 (10) | 3 (5)
Gait abnormal (General disorders) | 0 (0) | 1 (1) | 2 (2)
Hernia pain (General disorders) | 1 (1) | 2 (3) | 1 (2)
Inflammation localised (General disorders) | 2 (3) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 3 (7) | 8 (12) | 4 (6)
Infusion site pain (General disorders) | 3 (5) | 3 (3) | 2 (2)
Infusion site swelling (General disorders) | 4 (6) | 4 (4) | 1 (1)
Injection site bruising (General disorders) | 0 (0) | 2 (3) | 0 (0)
Injection site extravasation (General disorders) | 2 (2) | 2 (3) | 2 (3)
Injection site haemorrhage (General disorders) | 1 (1) | 0 (0) | 2 (2)
Lethargy (General disorders) | 2 (4) | 0 (0) | 0 (0)
Malaise (General disorders) | 5 (7) | 1 (1) | 3 (3)
Oedema peripheral (General disorders) | 2 (11) | 0 (0) | 1 (1)
Pain nos (General disorders) | 1 (1) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 20 (83) | 18 (68) | 19 (63)
Rigors (General disorders) | 1 (1) | 3 (8) | 1 (1)
Sensation of foreign body nos (General disorders) | 2 (2) | 0 (0) | 0 (0)
Ear infection nos (Infections and infestations) | 8 (15) | 9 (17) | 9 (19)
Furuncle (Infections and infestations) | 1 (1) | 2 (3) | 1 (1)
Herpes simplex (Infections and infestations) | 2 (2) | 1 (4) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 2 (2) | 3 (3)
Influenza (Infections and infestations) | 2 (2) | 1 (1) | 1 (2)
Lice infestation (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Localised infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Lower respiratory tract infection nos (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Otitis media nos (Infections and infestations) | 6 (8) | 7 (11) | 7 (9)
Otitis media serous nos (Infections and infestations) | 4 (8) | 2 (7) | 4 (6)
Respiratory tract infection nos (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Sinusitis nos (Infections and infestations) | 5 (5) | 2 (5) | 3 (4)
Tonsillitis (Infections and infestations) | 2 (2) | 3 (3) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1) | 1 (1) | 3 (4)
Upper respiratory tract infection nos (Infections and infestations) | 12 (26) | 12 (34) | 10 (19)
Urinary tract infection nos (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Varicella (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Viral infection nos (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Abrasion nos (Injury, poisoning and procedural complications) | 0 (0) | 3 (6) | 3 (6)
Arthropod bite (Injury, poisoning and procedural complications) | 3 (5) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 4 (5) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Post procedural pain (Injury, poisoning and procedural complications) | 2 (3) | 3 (5) | 3 (3)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 4 (6)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 3 (3)
Blood alkaline phosphatase nos increased (Investigations) | 1 (1) | 2 (2) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 2 (3) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Electrocardiogram abnormal nos (Investigations) | 1 (1) | 2 (2) | 0 (0)
Gamma-Glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (3)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Appetite decreased nos (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (26) | 14 (28) | 9 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (10) | 11 (25) | 8 (11)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4) | 0 (0)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (4) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (8) | 3 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 4 (4) | 3 (7)
Pain in foot (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (3) | 2 (2)
Pain in limb (Musculoskeletal and connective tissue disorders) | 9 (20) | 9 (18) | 10 (14)
Peripheral swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 2 (3)
Carpal tunnel syndrome (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 4 (10) | 6 (9) | 8 (16)
Headache (Nervous system disorders) | 19 (132) | 21 (118) | 14 (80)
Hyperreflexia (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Insomnia (Nervous system disorders) | 1 (1) | 3 (22) | 1 (3)
Migraine nos (Nervous system disorders) | 2 (2) | 0 (0) | 1 (3)
Paraesthesia (Nervous system disorders) | 2 (6) | 2 (2) | 1 (3)
Post-Traumatic headache (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1)
Tremor (Nervous system disorders) | 2 (4) | 1 (1) | 1 (1)
Abnormal behaviour nos (Psychiatric disorders) | 2 (2) | 0 (0) | 3 (3)
Anxiety (Psychiatric disorders) | 2 (4) | 4 (5) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
Asthma nos (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (3) | 2 (4)
Bronchitis nos (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Bronchospasm nos (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 2 (5) | 4 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (30) | 16 (38) | 19 (42)
Dyspnoea nos (Respiratory, thoracic and mediastinal disorders) | 4 (10) | 3 (3) | 9 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (5) | 4 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (4) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 12 (18) | 16 (39) | 12 (23)
Nasal passage irritation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 8 (16) | 5 (15)
Obstructive airways disorder nos (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 13 (19) | 11 (23) | 10 (18)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (3)
Rhinitis allergic nos (Respiratory, thoracic and mediastinal disorders) | 3 (7) | 3 (3) | 3 (6)
Rhinitis nos (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0) | 4 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9 (14) | 10 (19) | 9 (20)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 5 (9)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 3 (4)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 2 (3)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 5 (7) | 5 (8)
Acne nos (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 0 (0)
Contusion (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (6) | 2 (2)
Dyshidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 1 (2)
Erythema (Skin and subcutaneous tissue disorders) | 2 (12) | 1 (3) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (19) | 6 (14) | 5 (10)
Rash macular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Rash nos (Skin and subcutaneous tissue disorders) | 8 (14) | 11 (39) | 10 (29)
Rash pruritic (Skin and subcutaneous tissue disorders) | 5 (9) | 5 (6) | 0 (0)
Sweating increased (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2) | 3 (3)
Urticaria nos (Skin and subcutaneous tissue disorders) | 5 (10) | 4 (9) | 0 (0)
Flushing (Vascular disorders) | 5 (9) | 5 (9) | 6 (7)
Hypertension nos (Vascular disorders) | 8 (23) | 5 (7) | 7 (10)
Hypotension nos (Vascular disorders) | 3 (5) | 2 (4) | 4 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days